CLINICAL TRIAL: NCT02853565
Title: A Phase I Study of CAN008 Plus Concomitant Temozolomide During and After Radiation Therapy in Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: A Study of CAN008 for Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CANbridge Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN-B1-008-L-002
Record Dates: First submitted 2016-07-11; First posted 2016-08-03 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2017-09

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — APG101

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAN008 (Experimental): CAN008 administered as a 30 min intravenous infusion once a week until disease progression or unacceptable toxicity.
  Interventions: Drug: CAN008

INTERVENTIONS:
Drug: CAN008 — The dose escalation in the phase I study including 200mg in the first cohort and 400mg in the second cohort to Recommended for Phase 2 Dose (RP2D)
  Other Names: APG101

SUMMARY:
To evaluate CAN008 safety, tolerability, and pharmacokinetics (PK) of CAN008 when administered concurrent Plus Concomitant Temozolomide During and After Radiation Therapy in Patients with Newly Diagnosed Glioblastoma Multiforme.

DETAILED DESCRIPTION:
CAN008 is a glycosylated fusion protein consisting of the extracellular domain of human CD95 (APO-1/Fas) and the Fc domain of human IgG1. CAN008 blocks the interaction between CD95 and its cognate ligand CD95L. The target of CAN008 is the inhibition of CD95L. CD95L is expressed in glioblastoma whose cells are resistant to CD95-mediated apoptosis. CD95L was shown to be a crucial trigger in invasion and migration of tumor cells and neutralizing CD95L abolishes the invasive capacity of glioblastoma cells.

The purpose of the study is:

1. To describe the toxicity associated with this regimen in adult patients with newly diagnosed glioblastoma multiforme.
2. To determine the duration of disease free survival and overall survival associated with this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and histologically confirmed glioblastoma multiforme
* Tumor must be surgically accessible and tissue must be available
* Age ≥ 20 years and < 75 years
* Life expectancy ≥ 6 months
* Baseline MRI images must be done within 2 days after surgery
* Patients must have a Karnofsky performances score ≥ 60 prior to treatment.
* Patients must not have received prior cytotoxic drug therapy, non-cytotoxic drug therapy, or experimental drug therapy for brain tumors.
* Adequate hematologic (absolute neutrophil count (ANC) ≥ 1.5x109/L, platelet count ≥ 100x109/L, hemoglobin ≥ 10 g/dL ), renal (creatinine ≤ 1.25xULN ), and hepatic function (total bilirubin ≤ 1.5xULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5xULN)
* Women with childbearing potential must have a negative serum pregnancy test less than 7 days prior to the first dose of study drug.
* Both men and women of reproductive potential agree to use approved contraception, such as condom and placement of an intrauterine device (IUD), during the study and until 3 months after the discontinuation of study treatment.
* Willing and able to comply with the protocol as judged by the investigator
* Patients must provide written consent

Exclusion Criteria:

* Any prior chemotherapy (including carmustine-containing wafers) or immunotherapy (including vaccine therapy )
* Any prior radiotherapy to the brain
* Any concurrent malignancy other than basal cell carcinoma or carcinoma in situ of the cervix. Patients with a previous malignancy but without evidence of disease for ≥ 5 years will be allowed to enter the trial
* Any contraindication to TMZ listed in the local label
* Low-grade astrocytoma
* Unable to undergo MRI
* Past medical history of disease with poor prognosis according to the judgment of the Investigator
* HIV infection
* Patients with positive anti-HCV
* Patients with positive HbsAG who received any related treatment within the past 6 months
* Patients suffering from hereditary fructose intolerance (HFI).
* Patients receive any investigational agent(s) or device(s) within 30 days prior to entering the study
* Known coronary artery disease, significant arrhythmias or severe congestive heart failure

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 2 years
  The safety assessment will include safety laboratory (clinical chemistry, hematology, urinalysis), physical exam, vital signs and 12-lead ECG (QT prolongation). An AE can be any unfavourable and unintended sign, symptom, or disease temporarily associated with the use of a medicinal product, whether or not is considered to be related to the medicinal product. Pre-existing conditions worsen during a study are also to be reported as AEs. Furthermore, any side effects potentially related to the CAN008 treatment will be evaluated.

SECONDARY OUTCOMES:
Recommended Dose for Phase II [RP2D] measured by the Maximum Tolerated Dose [MTD] or the Maximum Administered Dose [MAD] | up to 2 years
  The RP2D will be determined based on the assessment of the observed toxicities, the maximum tolerated dose (MTD) or the maximum administered dose (MAD), and the overall safety profile of CAN008.
PK profile measured by CAN008 serum concentrations | up to 2 years
  CAN008 serum concentrations will be determined.
PK profile measured by Maximum Plasma Concentration [Cmax] | up to 2 years
  Maximum Plasma Concentration [Cmax] will be determined.
PK profile measured by Area Under the Curve [AUC] | up to 2 years
  Area Under the Curve [AUC] will be determined.
Preliminary efficacy (Progression Free Survival after 6 months [PFS6]) | up to 2 years
  PFS is defined as the time from date of randomization to the date of the event, which is the first radiologically documented disease progression (per local investigator assessment according to Response Assessment in Neuro-Oncology (RANO) criteria) or death due to any cause. For the primary analysis, progression-free survival after 6 months (PFS6) is defined as the crude rate of patients confirmed to be free of progression at 6 months after randomization with respect to the number of randomized and exposed patients in the respective treatment arm.
Preliminary efficacy (Overall Survival [OS]) | up to 2 years
  Overall survival (OS) is defined as the time from the first dose of CAN008 to death.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Xu, MD, Study Director — CANbridge Life Sciences Ltd.
Locations (2):
- Taiwan (2):
  - Chang Gung Memorial Hospital, Linkou, Taipei
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wei KC, Hsu PW, Tsai HC, Lin YJ, Chen KT, Toh CH, Huang HL, Jung SM, Tseng CK, Ke YX. Safety and tolerability of asunercept plus standard radiotherapy/temozolomide in Asian patients with newly-diagnosed glioblastoma: a phase I study. Sci Rep. 2021 Dec 15;11(1):24067. doi: 10.1038/s41598-021-02527-1. PMID 34911992